CLINICAL TRIAL: NCT03878433
Title: Oral Superoxide Dismutase (GLISODin) to Decrease Melasma Severity. A Prospective Randomized Placebo-controlled Study
Brief Title: Oral Superoxide Dismutase (GLISODin) to Decrease Melasma Severity.
Acronym: Glisodin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 18-PP-02
Record Dates: First submitted 2019-01-25; First posted 2019-03-18 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug (Active Comparator): Glisodin : 2 capsules of GliSODin, 500mg of GliSODIn per day. Preferably to take in the morning during breakfast
  Interventions: Drug: Glisodin
- No Drug (Placebo Comparator): 2 capsules of PLacebo, 500mg of Placebo per day. Preferably to take in the morning during breakfastbo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Glisodin — 500 mg/day between 12 weeks
  Arms: Drug
Other: placebo — Placebo group (20 patients) will receive 2 pills of placebo per day + sunscreen for 6 months
  Arms: No Drug

SUMMARY:
Oxidative stress has been reported to play a role in melasma pathophysiology. The objective of the study is to compare oral superoxide dismutase (GLISODin) to placebo, in combination to sunscreen to decrease melasma severity.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed melasma in adult patient
* signed inform consent

Exclusion Criteria:

* Pregnant women
* Other pigmentary disorder of the afce
* Use of depigmentant agent in the month before the inclusion
* Use of topical steroid, tretinoin, hydroquinone in the month before the inclusion
* Coeliac disease or allergy to gluten

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Severity of melasma | At baseline and at 12 weeks
  Change from Baseline of the Modified Melasma Area and Severity Index (mMASI) total score at 12 months. The MASI is 0 à 24 : Front 0.3(D)(A)+ right malar 0.30(D)(A)+ left malar 0.30(D)(A)+ chin 0.1(D)(A)

SECONDARY OUTCOMES:
Quality of life of patient: VAS (Visual Analog Scale) | At baseline and at 12 weeks
  Change from Baseline of quality of life at 12 months (Visual Analog Scale with a graduation from 0 to 10)
Satisfaction of the patients: VAS (Visual Analog Scale) | At baseline and at 12 weeks
  Change from Baseline of satisfaction of the patients total score at 12 months (Visual Analog Scale with a graduation from 0 to 10)

CONTACTS AND LOCATIONS:
Overall Officials: Passeron Thierry, PhD, Principal Investigator — Dermatologie, CHU de Nice
Locations (1):
- CHU de Nice - Dermatology, Nice, Alpes-Maritime, France

IPD SHARING:
Plan to Share IPD: No